CLINICAL TRIAL: NCT07097103
Title: A 2x2 Factorial Randomized Controlled Non-pharmacological Interventional Multicenter Pilot Study on the Influence of the Mediterranean Diet and Physical Exercise on the Microbiome of Patients With Parkinson's Disease
Brief Title: Parkinson's Research In Metagenomic Early Stage Biomarkers
Acronym: PRIME_2025
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: San Raffaele Cassino, Cassino, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RP 340/SR/25
Record Dates: First submitted 2025-06-30; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: Physical activity; Mediterranean Diet; Pilot study; Microbiome; Parkinson's disease
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: It's a 2x2 factorial, randomized, controlled, non-pharmacological intervention pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mediterranean Diet Intervention (Group A) (Experimental): Participants receive a structured Mediterranean Diet intervention, including personalized counseling, meal plans, educational sessions and monitoring.
  Interventions: Behavioral: Mediterranean Diet Intervention
- Intensive Physical Activity Intervention (Group B) (Experimental): Participants engage in a supervised structured physical activity program.
  Interventions: Behavioral: Intensive Physical Activity Intervention
- Mediterranean Diet + Intensive Physical Activity Combined Intervention (Group C=A+B) (Experimental): Participants will receive both dietary and physical activity interventions.
  Interventions: Behavioral: Mediterranean Diet Intervention; Behavioral: Intensive Physical Activity Intervention
- Controls (Group D) (Active Comparator): Participants continue their usual Parkinson's disease treatments according to clinical guidelines, without any additional specific dietary or exercise interventions provided by the study.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Mediterranean Diet Intervention — Participants will follow a personalized diet plan over 24 weeks, based on the guidelines of the Mediterranean diet and defined according to their needs and the state of the disease; no food category will be excluded a priori. Individualized nutritional counseling and support materials (weekly meal plans, sample recipes, portion guides) will be provided by a qualified nutritionist. Adherence to the Mediterranean diet will be monitored periodically. Participants will maintain their usual diet during a pre-baseline period of at least 4 weeks, then switch to the Mediterranean plan under the supervision of a nutritionist.
  Arms: Mediterranean Diet + Intensive Physical Activity Combined Intervention (Group C=A+B); Mediterranean Diet Intervention (Group A)
Behavioral: Intensive Physical Activity Intervention — Participants will perform exercise, over 24 weeks, according to WHO recommendations for adults, including those aged ≥ 64 years, to achieve at least 150-300 minutes of moderate-intensity aerobic physical activity, or at least 75-100 minutes of vigorous-intensity aerobic physical activity, or an equivalent combination of moderate and vigorous activity during the week. The WHO 2020 also recommend moderate-intensity or greater muscle-strengthening exercises involving alla major muscle groups for 2 or more days per week. Adherence will be monitored during in-person sessions and through wearable devices for activity tracking.
  Arms: Intensive Physical Activity Intervention (Group B); Mediterranean Diet + Intensive Physical Activity Combined Intervention (Group C=A+B)
Other: Control — Participants will continue their usual medical management for early Parkinson's disease according to current clinical guidelines, without any additional dietary or exercise interventions provided by the study, and will be monitored through standard follow-up visits but will not receive any study-specific dietary or physical activity programs.
  Arms: Controls (Group D)

SUMMARY:
This 2x2 factorial, randomized, controlled pilot study aims to identify a specific microbiota pattern, which could constitute a biomarker of Parkinson's disease, and to evaluate whether specific pathotypes can be associated with different stages of the disease; furthermore, the investigators are committed to evaluating how and to what extent the changes induced by a personalized nutritional intervention combined with physical exercise affect the symptoms and quality of life of patients.

DETAILED DESCRIPTION:
The study will last 60 months, and the following activities are planned:

* Study presentation, selection and enrollment of patients;
* Evaluation of patients' health and nutritional status, including collection of physiological, pathological, and pharmacological history;
* Randomization of patients into four groups;
* Sample collection and storage;
* Microbiome analysis;
* Evaluation of motor and non-motor symptoms using clinical tests and rating scales at baseline (T0), at six months (T1) after treatment initiation, and at three and six months post-intervention (FU1 and FU2, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to United Kingdom (UK) Parkinson's Disease Society Brain Bank criteria;
* aged 35-80 years;
* Hoehn & Yahr stage > 1 and < 3 in the clinical "ON" state;
* MoCA score ≥17.54;
* MMSE ≥24;
* Stable dopaminergic midication regimen for ≥ 4 weeks;
* Ability to interact with the research team and provide informed consent in Italian;
* Suitable to physical exercise;
* Able to walk unassisted (no walking aids);
* Willingness and ability to comply with all study procedures;
* Willingness to maintain usual diet during a ≥ 4-week pre-baseline period;
* Willingness to switch to a Mediterranean-style diet during the intervention;
* Ability to provide stool samples at each collection timepoint;
* Willing to avoid strenuous exercise and alcohol for 24 hours prior to each visits.

Exclusion Criteria:

* Pre-existing psychiatric disorders;
* Atypical or secondary Parkinsonism;
* Presence of pacemakers or other subcutaneous electronic devices;
* Any other neurological or neurodegenerative disorders;
* Moderate to severe cognitive decline;
* Beck Depression Inventory-II (BDI-II)] score ≥28;
* Dementia diagnosis;
* Thyroid dysfunctions;
* Type1 Diabetes Mellitus;
* Type 2 diabetes mellitus with HbA₁c ≥ 8% or on insulin therapy;
* Acute diseases;
* Active Neoplasia;
* IBD or IBS;
* Celiac disease;
* History of major gastrointestinal surgery or acute GI conditions (e.g., gastroenteritis) within the past 3-6 months;
* Chronic corticosteroid therapy;
* Use of proton pump inhibitors within the past 30 days;
* Acute, antibiotic-resistant infections;
* Antibiotic intake within the past 30 days;
* Prebiotic/probiotic supplement use in the past 30 days;
* Prolonged intake of anxiolytic drugs, antidepressants, antipsychotics, cognitive stimulants, and analogs in the past 3 months;
* Underweight (BMI <18.5);
* History of deep brain stimulation (DBS) surgery;
* Pregnancy or lactation;
* Regular use of enemas or suppositories to alleviate constipation;
* Use of experimental products in the 3 months prior to the screening visit
* Patients who, for medical reasons, are required to follow special dietary regimens that could interfere with the adoption or effectiveness of the Mediterranean model;
* Vegan/Vegetarian diet or any other dietary behaviour that excludes one or more of the typical food groups of the Mediterranean model.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-07-11 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Alpha Diversity of the fecal microbiota. | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in fecal microbiota alpha diversity, a measure of the richness and evenness of microbial species within a sample, will be assessed.
Beta Diversity of the fecal microbiota | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in fecal microbiota beta diversity, refers to the degree of difference in microbial community composition between different fecal samples, will be assessed.
Enterobacteriaceae species abundance across Parkinson's disease stage | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in fecal microbial composition will be assessed. Specifically, we will measure the relative abundance of Enterobacteriaceae species and pathotypes across different stages of Parkinson's disease.
Fecal Microbial relative quantification | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in relative quantification

SECONDARY OUTCOMES:
Intestinal Inflammation | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in fecal calprotectin (a valid and non-invasive marker of mucosal inflammation) will be assessed using enzyme-linked immunosorbent assay (ELISA).
Intestinal Permeability | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in fecal zonulin will be assessed using enzyme-linked immunosorbent assay (ELISA). The unit for measuring zonulin in stool samples is nanograms per milliliter (ng/mL). The Protein Zonulin is a very important indicator for leaky gut.
Changes in extracellular vesicle concentration (particles/mL) in saliva and plasma will be assessed. | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  To evaluate the effect of the combined diet and physical activity intervention on extracellular vesicles (EVs), EVs will be isolated from saliva and plasma by serial ultracentrifugation and size-exclusion chromatography. EV concentration and size distribution will be determined by nanoparticle tracking analysis (NTA).
Changes in protein marker expression in saliva and plasma. | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Extracellular Vesicles (EVs)-associated proteins (CD63, CD9, α-synuclein, BDNF, L1CAM, and CD56) will be quantified by dot blot and confirmed by fluorescent NTA and/or cytofluorimetric analysis.

OTHER OUTCOMES:
Total score on the Digestion-Associated Quality of Life Questionnaire (DQLQ) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Participants will complete the Digestion-Associated Quality of Life Questionnaire (DQLQ) for a total of 9 statements. Possible totale score ranges from 0 to 9, with a higher score indicates a lower (worse) digestion-associated QoL
Changes in non-motor symptoms MDS-UPDRS Part I | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I (non-motor symptoms of daily living) scores will be assessed. The minimum score on the MDS-UPDRS Part I is 0 and the maximum is 52, with higher scores representing worse non-motor symptoms of daily living.
Changes in motor symptoms MDS-UPDRS Part II | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II (motor symptoms of daily living) scores will be assessed. The minimum score on the MDS-UPDRS Part II is 0 and the maximum is 52, with higher scores representing worse motor symptoms of daily living.
Changes in motor symptoms MDS-UPDRS Part III | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II (motor examination) scores will be assessed. The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132, with higher scores representing worse motor symptoms.
Changes in motor symptoms MDS-UPDRS Part IV | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV (motor complications) scores will be assessed. The minimum score on the MDS-UPDRS Part IV is 0 and the maximum is 24, with higher scores representing worse motor complications.
Changes in motor symptoms (H&Y) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in The Hoehn & Yahr scale (H&Y) scale will be assessed. H&Y scale is a system used to describe the progression of motor symptoms in PD - it ranges from Stage 0 (no signs of disease) to Stage 5 (wheelchair-bound or bedridden).
Changes in movement analysis (TUG) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in the execution time of the Timed Up & Go (TUG) test-a reliable and valid measure of mobility, balance, walking ability, and fall risk-will be assessed.
Change in postural instability | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Berg Balance Scale (BBS), a 14-item objective measure that assesses static balance and fall risk in adults. Each item is scored on a 5-point ordinal scale ranging from 0 to 4, with 0 indicating an inability to complete the task entirely and 4 indicating an ability to independent complete the task ,
Change in movement analysis - propulsion | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in propulsion (anterior-posterior peak acceleration during the lower-limb swing phase, measured by a wearable G-sensor in m/s²) will be assessed.
Change in walking capacity | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in the 10-Meter Walking Test, a standardized method used to assess gait speed and functional mobility.
Changes in Gastrointestinal symptoms | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in "Gastrointestinal Symptom Rating Scale" (GSRS), a specific tool consisting of 15 items, that are grouped into five symptom clusters: reflux, abdominal pain, indigestion, diarrhea, constipation.
Changes in stool types | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Bristol Stool Scale, a diagnostic medical tool designed to classify the form of human faeces into seven categories (Type 1 and 2: May be difficult to pass, may indicate constipation; Type 3 and 4: Ideal stools; Type 5: Trending toward diarrhea; Type 6 and 7: Diarrhea).
Change in non-motor symptoms (NMSS) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Non-motor Symptom Scale (NMSS), a 30-item scale including the following 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems, attention/memory, gastrointestinal, urinary, sexual function and miscellaneous.
Changes in severity of depressive symptomatology | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Beck Depression Inventory-II (BDI-II), a 21-item self-report inventory measuring the severity of depression.
Changes in quality of life | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Parkinson's Disease Questionnaire-39 (PDQ-39), a tool assessing QoL in eight domains (mobility, daily activities, emotional well-being, stigma, social support, knowledge, communication, and physical discomfort). It's a 5-point scale for each of the 39 questions (0=Never; 1=Rarely; 2=Sometimes; 3=Often; 4=Always). The minimum score is 0 means good health, maximum score is 100 means bad health; a higher score indicates a lower QoL.
Changes in cognitive function - Mini-Mental State Examination (MMSE) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Mini-Mental State Examination (MMSE), a 30-point items to measure cognitive impairment examining functions like registration, attention and calculation, recall, language, ability to follow simple commands and orientation.
Change in cognitive function - Montreal Cognitive Assessment (MoCA) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Montreal Cognitive Assessment (MoCA), a 10-minute test used to detect cognitive impairment related to PD.
Change in cognitive function - Frontal Assessment Battery (FAB) | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)
  Changes in Frontal Assessment Battery (FAB), a 10 minutes tool evaluating the executive functions located in the frontal lobes, consisting of 6 tests that correspond to each specific cognitive or behavioral domain related to the frontal lobes; FAB scores range between 0 and 18, with higher scores representing a better outcome.
Changes in cognitive abilities | Baseline (Week 0); End of intervention (Week 24); First Follow-up (Week 36); Second Follow-up (Week 48)Chan
  Changes in Clock Drawing Test, a simple tool used to check for signs of dementia, that measures several cognitive abilities at once, including attention, hearing comprehension, visual memory, and motor skills.

IPD SHARING:
Plan to Share IPD: No